CLINICAL TRIAL: NCT02519569
Title: Internet-based Intervention for Complicated Grief: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Tromso (Other)
Responsible Party: Principal Investigator, Jens Thimm, Associate professor, University of Tromso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/388(REK)
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Complicated Grief

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): Internet-based cognitive-behavioral therapy for complicated grief
  Interventions: Other: Internet-based cognitive-behavioral therapy

INTERVENTIONS:
Other: Internet-based cognitive-behavioral therapy — The intervention consists of ten writing assignments

SUMMARY:
A considerable proportion of bereaved individuals experience chronic and disabling grief (so-called complicated or prolonged grief). Complicated grief is associated with severe mental and physical health problems as well as impaired social and occupational functioning. Interventions based on cognitive-behavioral therapy and applied via the internet have shown to be efficacious for this condition, but have not yet been adapted and evaluated in Norway. The aim of the current study is to adapt an internet-based cognitive-behavioral intervention for complicated grief and evaluate its effectiveness as a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Complicated grief
* Internet access
* Fluent in Norwegian
* No concomitant psychological treatment

Exclusion Criteria:

* Severe depression
* Psychotic symptoms
* Dissociation
* Suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from pretest to posttest in symptoms of complicated grief | 6 weeks
Change from pretest to follow-up (1) in symptoms of complicated grief | 18 weeks
Change from pretest to follow-up (2) in symptoms of complicated grief | 30 weeks

SECONDARY OUTCOMES:
Change from pretest to posttest in posttraumatic growth | 6 weeks
Change from pretest to follow-up (1) in posttraumatic growth | 18 weeks
Change from pretest to follow-up (2) in posttraumatic growth | 30 weeks
Change from pretest to posttest in quality of life | 6 weeks
Change from pretest to follow-up (1) in quality of life | 18 weeks
Change from pretest to follow-up (2) in quality of life | 30 weeks
Change from pretest to posttest in depression | 6 weeks
Change from pretest to follow-up (1) in depression | 18 weeks
Change from pretest to follow-up (2) in depression | 30 weeks